CLINICAL TRIAL: NCT03448614
Title: Skull Base Reconstruction After Endonasal Cranio-endoscopic Resection Using Autologus Grafts
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Sholkamy, dr, Assiut University
Other Study IDs: skull base reconstruction
Record Dates: First submitted 2018-01-06; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Skull Base Neoplasms
Keywords: skull base reconstrction
MeSH Terms: conditions — Skull Base Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endonasal endoscopic approach to the skull base has been expanded in the last several years owing to advances in the radiological aspect that provided a better evaluation of the lesions and the surrounding structures, technological advances that include angled endoscope, development of high-resolution cameras, high definition monitors and navigation systems and better anatomical experience. The endoscopic endonasal approach now provides access to frontal sinus to the second cervical vertebra in the sagittal plane and from the sella to the jugular foramen in the coronal plane. Endoscopic resection of large skull base tumors results in large defect for which repair is a challenge. Several factors besides the size of the defect should be considered during skull base repair as CSF leak, CSF pressure, history or need for future radiotherapy, lack of support and local tissue vascularity. The aim of this study is to Provide an algorithmic approach for skull base reconstruction after endonasal cranio-endoscopic resection using autologous grafts according to the extent of resection, skull base defect size, the presence of CSF leak, CSF pressure and local tissue vascular

DETAILED DESCRIPTION:
Type of the study:

A prospective clinical study will be conducted in the period between January 2018 and January 2020.

Study Setting:

Otolaryngology Department, Alexandria University Hospital. Otolaryngology Department, Assiut University Hospital.

Study tools :

Preoperative evaluation:

1. Personal history: age, sex, marital status, occupation, number of children, and endocrinal history in case pituitary tumors.
2. Presentation: endocrine, visual, oculomotor and/or a headache.
3. Therapeutic history.
4. Past history: trans-sphenoidal surgery, trauma and nasal diseases and/or surgery.
5. General examination: including gross features of Cushing's disease or acromegaly.
6. Full ENT examination including assessment of the nasal cavity, nasal septum for deviation, perforation and/or adhesions) and nasal turbinates; including nasal endoscopic examination and dental assessment.
7. Neurosurgical consultation.
8. Ophthalmological assessment: visual acuity, visual field, fundus examination and color vision.
9. Radiological assessment:

   1. MRI of the brain: A complete protocol including at least, T1- and T2-weighted images and T1-weighted post-contrast (gadolinium) images, in the three orthogonal planes at max 3 mm sections: for assessment of tumor site, size and extension, and involvement of large blood vessels and nerves.
   2. Multi-slice CT scan of the nose and paranasal sinuses (bone window, high resolution, with intravenous contrast, in the three orthogonal planes, with three-dimensional reconstruction and at maximum 3 mm sections): for assessment of nasal cavity abnormalities including the nasal septum, sinus pathology, type of sphenoid sinus pneumatization, etc.
10. Assessment of the general condition of the patient:

    1. Complete blood count: to assess for anemia or other hematological abnormalities.
    2. Serum electrolytes: mainly sodium and potassium.
    3. Fasting and postprandial blood glucose level.
    4. ECG and echocardiography.

Operative techniques:

After cranio-endoscopic resection and complete removal of the lesion skull base defect will be repaired according to the following scheme (modified from Sigler et al) No leak →No repair or single layer Low-flow leak → Multilayer repair Autograft (fascia Lata, fat, bone, mucosa) High-flow leak →Multilayer repair Autograft (fascia Lata, fat, bone, mucosa)+ Intranasal vascularized flap.

Modifying factors (factors that indicate the need for a vascularized flap regardless of leak type): Cushing disease, morbid obesity, craniopharyngioma, meningioma, extended skull base approach, large defect, revision surgery, history of or future need for radiation treatment.

So repair technique after extensive dural and bony resection or high flow leak will include multiple layers of fascia lata with pieces of fatty tissue in between. After that, a nasoseptal flap (or other vascularized flap, e.g., posterior pedicled inferior turbinate, posterior pedicled middle turbinate, bipedicled anterior septal, anterior inferior turbinate) will be harvested and applied according to local vascularity.

Then a separator will be applied; to prevent future accidental dislodgement of grafts during Merocel® removal, followed by placement of a moderately inflated Foley balloon catheter; to support the reconstruction.

At the end of the procedure, when hemostasis will be achieved, irrigation will be performed to remove any bone residuals or blood clots from the choanae and the nasopharynx. Then, the middle turbinates will be gently repositioned medially. At last, nasal Merocel® (polyvinyl alcohol) sponges will be placed in the nasal cavity on either side and hydrated with saline to expand.

Repair of low flow leak will be the same as the previous technique with the replacement of the vascularized flap with free mucosal graft and no need for Foley catheter.

Early postoperative management:

For the next twenty-four hours, the patient will be monitored in the intensive care unit, particularly for diabetes insipidus (after pituitary surgery), visual deterioration, any CSF leak, manifestations of meningitis or any hemorrhage.

Inspection for CSF leak will be a part of the routine evaluation of every patient, both in the recovery room and in the days after surgery. If persistent CSF leak became evident, a lumbar drainage was tried before re-exploration under general anesthesia. Analgesics will be routinely prescribed. Prophylaxis against postoperative nausea and vomiting will be achieved by an intraoperative intravenous administration of a single dose of an antiemetic, ondansetron 4 mg, as well as a throat pack to prevent intraoperative bleeding from draining into the stomach.

An intravenous third-generation cephalosporin will be started with anesthesia induction and continued until removal of the nasal packing. Then, patients will be kept on a five days course of an oral antibiotic; for safety.

Nasal packs will be removed on the third or fifth postoperative day. Then, the patient will be examined under endoscopic guidance.

Follow up:

I. Otorhinolaryngologic assessment: The first office visit will be scheduled after a week following the surgery. After application of topical anesthesia (lidocaine 10%), any blood clots will be endoscopically removed and any synechiae will be released. The examination will be for any bleeding or CSF leakage. The patient will be seen on a weekly basis for the first three weeks and then every three weeks for the next two appointments. Healing usually occurs three to six weeks. Further appointments will be scheduled as necessary II. Neuro-radiological assessment: Early MRI will be obtained on the first or second postoperative day to assess the extent of resection, the location of the fat graft if one is present, and the presence of any hematoma. Serial imaging was done after six months and then annually.

III. Endocrinal assessment: in case of hypophysectomy. IV. Ophthalmological assessment: serial visual field, visual acuity, and fundus examinations will be done for every patient, especially those with a pre-operative visual loss.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing endonasal cranio-endoscopic resection

Exclusion Criteria:

* Unfit patient for surgery.
* Patient refusal to participate in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patient will undergo endonasal cranio-endoscopic resection
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Head CT scan | within 1month preoperative
  bone window axial, coronal and sagittal cuts to measure preoperative skull base defect size
brain MRI: with and without contrast | within1 week post operative
  Coronal, axial and sagittal MRI in T1 and T2 signals measures postoperative tumor, to assess the repaired defect after the surgery
brain MRI: with and without contrast | 3 monthes post operative
  Coronal, axial and sagittal MRI in T1 and T2 signals to assess the repaired defect after the surgery
brain MRI: with and without contrast | 6monthes postoperative
  Coronal, axial and sagittal MRI in T1 and T2 signals to assess the repaired defect after the surgery, recurrence of tumor

SECONDARY OUTCOMES:
estimation of incidence of sinonasal, orbital &/or intracranial complications | within 90 days following surgery
  identification of possible complication that will occur during resection of skull base and removal of tumors
the incidence of CSF leakage | within 90 days postoperative
  history of CSF leakage confirmed by endoscopic examination
CSF leakage related surgical intervention | within 90 days postoperative
  second surgical intervention to explore the grafted defect
Endonasal endoscopic evaluation of the grafted defect | within 1 month postoperative, 3monthes postoperative
  using 4 mm 0-degree endoscope to measure graft condition and visualize any CSF fistula
Brain MRI: with and without contrast | within 1 month preoperative
  Coronal, axial and sagittal MRI in T1 and T2 signals measures preoperative tumor size
type of pathology | within 1 week post operative
  identification of the type of the pathology

CONTACTS AND LOCATIONS:
Overall Officials: ahmed G sholkamy, Msc, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Kassam A, Snyderman CH, Mintz A, Gardner P, Carrau RL. Expanded endonasal approach: the rostrocaudal axis. Part I. Crista galli to the sella turcica. Neurosurg Focus. 2005 Jul 15;19(1):E3. PMID 16078817
- [Background] Kassam A, Snyderman CH, Mintz A, Gardner P, Carrau RL. Expanded endonasal approach: the rostrocaudal axis. Part II. Posterior clinoids to the foramen magnum. Neurosurg Focus. 2005 Jul 15;19(1):E4. PMID 16078818
- [Background] Kassam AB, Gardner P, Snyderman C, Mintz A, Carrau R. Expanded endonasal approach: fully endoscopic, completely transnasal approach to the middle third of the clivus, petrous bone, middle cranial fossa, and infratemporal fossa. Neurosurg Focus. 2005 Jul 15;19(1):E6. PMID 16078820
- [Background] Kassam A, Carrau RL, Snyderman CH, Gardner P, Mintz A. Evolution of reconstructive techniques following endoscopic expanded endonasal approaches. Neurosurg Focus. 2005 Jul 15;19(1):E8. PMID 16078822
- [Background] Snyderman CH, Kassam AB, Carrau R, Mintz A. Endoscopic Reconstruction of Cranial Base Defects following Endonasal Skull Base Surgery. Skull Base. 2007 Feb;17(1):73-8. doi: 10.1055/s-2006-959337. PMID 17603646
- [Background] Sigler AC, D'Anza B, Lobo BC, Woodard TD, Recinos PF, Sindwani R. Endoscopic Skull Base Reconstruction: An Evolution of Materials and Methods. Otolaryngol Clin North Am. 2017 Jun;50(3):643-653. doi: 10.1016/j.otc.2017.01.015. Epub 2017 Mar 31. PMID 28372814
- [Background] Villaret AB, Schreiber A, Battaglia P, Bignami M. Endoscopy-assisted iliotibial tract harvesting for skull base reconstruction: feasibility on a cadaveric model. Skull Base. 2011 May;21(3):185-8. doi: 10.1055/s-0031-1275260. PMID 22451823
- [Background] Zanation AM, Thorp BD, Parmar P, Harvey RJ. Reconstructive options for endoscopic skull base surgery. Otolaryngol Clin North Am. 2011 Oct;44(5):1201-22. doi: 10.1016/j.otc.2011.06.016. PMID 21978902
- [Background] Hadad G, Bassagasteguy L, Carrau RL, Mataza JC, Kassam A, Snyderman CH, Mintz A. A novel reconstructive technique after endoscopic expanded endonasal approaches: vascular pedicle nasoseptal flap. Laryngoscope. 2006 Oct;116(10):1882-6. doi: 10.1097/01.mlg.0000234933.37779.e4. PMID 17003708
- [Background] El-Sayed IH, Roediger FC, Goldberg AN, Parsa AT, McDermott MW. Endoscopic reconstruction of skull base defects with the nasal septal flap. Skull Base. 2008 Nov;18(6):385-94. doi: 10.1055/s-0028-1096202. PMID 19412408